CLINICAL TRIAL: NCT02600936
Title: Sinai Vein Stent Registry
Status: Recruiting | Type: Observational
Sponsor: Windsor Ting (Other)
Responsible Party: Sponsor-Investigator, Windsor Ting, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: GCO 14-1497
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Venous Outflow Obstruction
Keywords: venous outflow obstruction; peripheral venous disease; vein stent; Wallstent; registry; May Thurner

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Registry: A retrospective and prospectively maintained registry of patients who have undergone or will undergo vein stent placement for proximal venous outflow obstruction
  Interventions: Device: vein stent placement

INTERVENTIONS:
Device: vein stent placement — Venous outflow obstruction will be treated by the placement of a stent to keep the vein open. This procedure is a minimally invasive endovascular treatment.

SUMMARY:
The Sinai Vein Stent Registry aims to establish and maintain a registry of patients who have undergone a vein stent placement procedure at The Mount Sinai Medical Center. The purpose of this study is to monitor and evaluate the long-term outcomes of venous stents placed to treat venous outflow obstruction. Outcome variables that will be assessed are: patency rate, reintervention rate, occurrence of any complications, clinical improvement, and quality of life. Venous outflow obstruction is defined as a stenosis and/or occlusion seen primarily in the ilio-femoral vein and inferior vena cava, and infrequently in the subclavian vein, brachiocephalic vein, or superior vena cava. While vein stent placement procedures are currently being performed in the United States, using stents which are commercially available and FDA-approved for use in arterial interventions, at this time there are no stents that are FDA-approved for use in veins. The placement of stents in veins holds tremendous promise as a treatment for venous outflow obstruction, but review of current literature has showed a paucity of published data on the long-term outcomes of this treatment.

The study is composed of two arms, a retrospective arm and a prospective arm. Any patient over the age of 18 who has undergone or is scheduled to undergo a vein stent placement procedure is eligible for this study. A HIPAA waiver and waiver of informed consent are being requested for the retrospective arm for patients who have undergone a vein stent placement procedure from January 1st 2012 to date of study onset, as it is not possible to contact all patients in the retrospective arm (i.e., lost to follow-up, no longer follows-up with a study physician). This study is only interested in the collection and analysis of data; the clinical care and outcomes of research subjects will not be affected by their participation in this study.

An IDE application has been submitted to the FDA for use of the Wallstent™ (manufactured by Boston Scientific, Inc.) in veins as treatment for venous outflow obstruction. The primary stents being used as treatment for venous outflow obstruction at Mount Sinai is the Wallstent™, mainly due to the fact that only Wallstents™ are available in the appropriate sizes to be used in veins. In rare occasions or exceptional circumstances, a smaller self-expanding nitinol stent may be used. Due to the extremely rare frequency of stents other than Wallstents™ being used and the impracticality (if not impossibility) of obtaining IDEs for all other stents, the investigators believe it is appropriate to exclude usage of these stents from the study data. To confirm, the purpose of this study is to monitor and evaluate long-term outcomes of the venous stents/the vein stent placement procedure, not specifically the Wallstent™ itself.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient has undergone or will undergo vein stent placement for proximal venous outflow obstruction in the ilio-femoral vein, inferior vena cava, subclavian vein, brachiocephalic vein, or superior vena cava.

Exclusion Criteria:

* Patient declines participation in the study.
* Confirmed ipsilateral acute DVT of the iliac vein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient has undergone or will undergo vein stent placement for proximal venous outflow obstruction in the ilio-femoral vein, inferior vena cava, subclavian vein, brachiocephalic vein, or superior vena cava.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
lumen area of stent | 12 month
  change in lumen area of 50% or greater in diseased segment compared to maximal reference lumen area of stent as measured by venogram and/or intravascular ultrasound (IVUS)
stent occlusion | 12 month
  occlusion of any stent segment, either the entire stent or any segment of the implanted stent

SECONDARY OUTCOMES:
major adverse event occurrence | 30 day
  performance goal estimated at 1% or less. Major adverse events are defined as: 1) Death, by any cause, 2) Bleeding requiring surgical or endovascular intervention or blood transfusion >= 2 units that is considered probably or definitely related to the index procedure or device, 3) Vascular injury requiring surgical/endovascular intervention, 4) Clinically significant pulmonary embolism requiring anticoagulation and/or thrombolysis, 5) Embolization/migration of stent
reintervention rate | 12 month
  estimated at 10%.
Venous clinical severity score (VCSS) | 1 year
  The VCSS was developed from elements of the CEAP classification (clinical grade, etiology, anatomy, pathophysiology), which is the worldwide standard for describing the clinical features of chronic venous disease. Components rated 0-3, with 3 being severe.
VCSS | 3 years
  The VCSS was developed from elements of the CEAP classification (clinical grade, etiology, anatomy, pathophysiology), which is the worldwide standard for describing the clinical features of chronic venous disease. Components rated 0-3, with 3 being severe.
VCSS | 5 years
  The VCSS was developed from elements of the CEAP classification (clinical grade, etiology, anatomy, pathophysiology), which is the worldwide standard for describing the clinical features of chronic venous disease. Components rated 0-3, with 3 being severe.
CEAP score | 1 year
  Assess clinical improvement with CEAP, scored from 1-6 with 6 being severe (C- clinical manifestation E- etiologic factors A- anatomic distribution P- pathophysiologic dysfunction)
CEAP score | 3 year
  Assess clinical improvement with CEAP, scored from 1-6 with 6 being severe (C- clinical manifestation E- etiologic factors A- anatomic distribution P- pathophysiologic dysfunction)
CEAP score | 5 years
  Assess clinical improvement with CEAP, scored from 1-6 with 6 being severe (C- clinical manifestation E- etiologic factors A- anatomic distribution P- pathophysiologic dysfunction)

CONTACTS AND LOCATIONS:
Overall Officials: Windsor Ting, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Neglen P, Thrasher TL, Raju S. Venous outflow obstruction: An underestimated contributor to chronic venous disease. J Vasc Surg. 2003 Nov;38(5):879-85. doi: 10.1016/s0741-5214(03)01020-6. PMID 14603188
- [Background] Neglen P, Hollis KC, Olivier J, Raju S. Stenting of the venous outflow in chronic venous disease: long-term stent-related outcome, clinical, and hemodynamic result. J Vasc Surg. 2007 Nov;46(5):979-990. doi: 10.1016/j.jvs.2007.06.046. PMID 17980284
- [Background] Ye K, Lu X, Li W, Huang Y, Huang X, Lu M, Jiang M. Long-term outcomes of stent placement for symptomatic nonthrombotic iliac vein compression lesions in chronic venous disease. J Vasc Interv Radiol. 2012 Apr;23(4):497-502. doi: 10.1016/j.jvir.2011.12.021. Epub 2012 Feb 17. PMID 22342482
- [Background] O'Sullivan GJ, Sheehan J, Lohan D, McCann-Brown JA. Iliofemoral venous stenting extending into the femoral region: initial clinical experience with the purpose-designed Zilver Vena stent. J Cardiovasc Surg (Torino). 2013 Apr;54(2):255-61. PMID 23558660
- [Background] Raju S, Ward M Jr, Kirk O. A modification of iliac vein stent technique. Ann Vasc Surg. 2014 Aug;28(6):1485-92. doi: 10.1016/j.avsg.2014.02.026. Epub 2014 Mar 12. PMID 24632315